CLINICAL TRIAL: NCT06047236
Title: Immune Biomarker Study for Salivary Gland Carcinoma
Acronym: ImmoGlandula
Status: Recruiting | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: ImmoGlandula
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-09

CONDITIONS: Salivary Gland Tumor; Benign Salivary Gland Tumor
MeSH Terms: conditions — Salivary Gland Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In this study, the prognostic value of local immunological tumor-dependent cell populations will be prospectively investigated and correlated with immunological changes in the blood. Not only single immune cell populations but also the immune score of multiple immune cells or immune cell subsets will be investigated. In addition, the systemic immune status of patients in peripheral blood will be studied longitudinally. Furthermore, the analysis of cytokines and chemokines as well as mRNA and ctDNA in the peripheral blood is blood and the determination of transcription processes in immune cells, especially to extend the especially to extend the prognostic immune signature.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Observational Arm: Initial diagnosis of primary salivary gland carcinoma in the head and neck region
  Interventions: Other: Sampling
- Control Group 1: Initial diagnosis of a benign salivary gland tumor in the head and neck region
  Interventions: Other: Sampling
- Control Group 2: Healthy control group. Functional diseases of the nose or ear (patients with the indication for functional ear surgery and rhinoplasty) without salivary gland tumor.
  Interventions: Other: Sampling

INTERVENTIONS:
Other: Sampling — Evaluation of immune characteristics by using patient's stool, saliva and blood samples.

SUMMARY:
Aims of this study are analyses of tumor metabolome, tumor transcriptome and tumor proteome as well as of the immune infiltration, separated by histological entity. These data will subsequently be compared with the with the detailed immune status determined in the patient's peripheral blood and saliva using machine learning techniques, among others, to create a biomarker cluster for salivary gland tumors. These can be used in clinical routine.

In addition, the investigators would like to study a subset of patients from freshly resected tumor organoids from freshly resected tumor tissue according to already established methods in order to mechanistic investigations of prognostic parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Observational group

   * Initial diagnosis of a primary salivary gland carcinoma in the head and neck region (no squamous cell carcinomas)
   * Specimen collection from the center of the tumor when the primary tumor is sufficiently large without that the pathological assessment is impaired
2. Control group 1

   * Initial diagnosis of a benign salivary gland tumor in the head and neck region
   * Specimen collection from the center of the tumor when the primary tumor is sufficiently large without that the pathological assessment is impaired
3. Control group 2

   * functional diseases of the nose or ear (patients with the indication for functional ear surgery and rhinoplasty)
   * Specimen collection with sufficiently large resectate during a functional nose surgery

for all groups:

* Willingness of patients to collect blood, saliva and stool and consent to the preservation of all samples for study purposes.
* Age ≥ 18 years
* sufficient cognitive ability of the patients to understand the purpose of the study and to understand the purpose of the study and agree to it

Exclusion Criteria:

* Distant metastasis at the time of diagnosis and simultaneous second cancers, i.e. at study inclusion
* Malignancy in the last 5 years regardless of location (except basal cell carcinoma or cis of the uterine cervix)
* Carcinomas for which specimen collection is not possible or likely without compromising the compromise the pathological evaluation
* Persistent drug or medication abuse
* Patients who are unable or unwilling to comply with protocol and to be treated
* Patients who are represented by a legal guardian
* Patients who are not suitable for participation in the study due to a language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for treatment at the participating study centers and meeting the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Observation of changes in an established immune matrix (intratumoral and systemic) | Change of the immune matrix from baseline to the end of study period, up to 5 years
  Different immune cells and tumor cell markers will characterize immunological groups using cluster analysis. Immune matrix of patients assessed by liquid immune profile-based signature (LIPS) (acc. Zhou et al. Journal for ImmunoTherapy of Cancer (JITC), 2021) and Tumour Associated Lymphocytes (TAL).
Longitudinal immunophenotyping of the patients: Detection of about 30 distinct immune cell (sub)types together with their activation markers during study period | Change of the immunophenotyping from baseline to the end of study period, up to 5 years
  The distribution of immune cells and messenger substances in the blood will be examined by means of immunophenotyping in order to add the systemic immune cell composition.
  Flow cytometric assessment of the amount of circulating immune cell-distribution per milliliter whole blood according to the LIPS technique (Zhou et al. JITC 2021).
Analysis of cytokines in peripheral blood and their change at certain points in the course of treatment | Change of the cytokine expression from baseline to the end of study period, up to 5 years
  Electrochemiluminescent MULTI-ARRAY measurement of concentration (pg/ml whole blood) cytokines/chemoattractant cytokines in the serum/plasma of the patients according to the LIPS technique (Zhou et al. JITC 2021).
Analysis of patient's metabolic state | The analyses are conducted from baseline to the end of study period, up to 5 years
  Mass-spectrometric untargeted metabolomic of patients serum/plasma to assess the change of metabolites (pg/ml whole blood) from baseline to end of radiotherapy.
Analysis of patient's microbiomic state by examination of saliva, tumor and stool | The analyses are conducted from baseline to the end of study period, up to 5 years
  16S rRNA deep sequencing of microbiome in salvia, tumour and stool samples to assess the presence and relative distribution of microbiotes (Operational taxonomic units (OTUs)).

CONTACTS AND LOCATIONS:
Overall Officials: Sarina Mueller, PD, Study Director — Universitätsklinikum Erlangen, HNO; Marlen Haderlein, PD, Study Director — Universitätsklinikum Erlangen, Radiation Oncology; Benjamin Frey, PD, Principal Investigator — Universitätsklinikum Erlangen, Radiation Oncology, Translational Radiobiology
Locations (2):
- Germany (2):
  - Universitätsklinikum Erlangen, HNO, Erlangen, Bavaria
  - Universitätsklinikum Erlangen, Strahlenklinik, Erlangen, Bavaria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Donaubauer AJ, Frey B, Agaimy A, Lange F, Mogge L, Fietkau R, Iro H, Munoz LE, Weber M, Kesting M, Gaipl US, Haderlein M, Muller S. Definition of predictive and prognostic immune biomarkers for salivary gland cancer from the intratumoural and systemic immune status: detailed protocol of the prospective, observatory ImmoGlandula study. BMJ Open. 2026 Jan 12;16(1):e100021. doi: 10.1136/bmjopen-2025-100021. PMID 41526019